CLINICAL TRIAL: NCT06497556
Title: A Phase III, Randomized, Open-Label, Multicenter Study Evaluating the Efficacy and Safety of Divarasib Versus Sotorasib or Adagrasib in Patients With Previously Treated KRAS G12C-Positive Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Divarasib Versus Sotorasib or Adagrasib in Participants With Previously Treated KRAS G12C-positive Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: Krascendo 1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO45217; 2024-510908-37-00 (Other: EU CT Number)
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; KRAS G12C Lung Cancer
Keywords: Advanced Non-Small Cell Lung Cancer; KRAS G12 Lung Cancer; Advanced Lung Cancer; Metastatic lung cancer; Divarasib; KRAS G12C Inhibitor; KRAS G12C Positive; KRAS Mutation; KRAS G12C Mutation; Lung Cancer Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — sotorasib; adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Divarasib (Experimental): Participants will receive divarasib orally, once daily (QD).
  Interventions: Drug: Divarasib
- KRAS G12C inhibitor (Active Comparator): Participants will receive sotorasib orally QD or adagrasib orally twice a day (BID)
  Interventions: Drug: Sotorasib; Drug: Adagrasib

INTERVENTIONS:
Drug: Divarasib — Divarasib will be administered orally QD
  Arms: Divarasib
Drug: Sotorasib — Sotorasib will be administered orally QD
  Arms: KRAS G12C inhibitor
Drug: Adagrasib — Adagrasib will be administred orally BID
  Arms: KRAS G12C inhibitor

SUMMARY:
The purpose of this study is to assess the safety and efficacy of divarasib compared to locally approved KRAS G12C inhibitors (sotorasib or adagrasib) in participants with KRAS G12C-positive (KRAS G12C +) advanced or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal histologically or cytologically confirmed diagnosis of metastatic or locally advanced NSCLC not amenable to treatment with surgical resection or combined chemoradiation
* Disease progression during or after treatment with at least one prior systemic therapy but no more than three lines of prior systemic therapy in the advanced or metastatic setting
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Documentation of the presence of a KRAS G12C mutation
* Availability of a representative formalin-fixed, paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or 10-15 (15 preferred) unstained, freshly cut, serial slides with an associated pathology report
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of >= 12 weeks

Exclusion Criteria:

* Known hypersensitivity to any of the components of divarasib, or sotorasib or adagrasib
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Known concomitant second oncogenic driver
* Mixed small-cell lung cancer or large cell neuroendocrine histology
* Known and untreated, or active central nervous system (CNS) metastases
* Leptomeningeal disease or carcinomatous meningitis
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures biweekly or more frequently
* Any infection that, in the opinion of the investigator, could impact patient safety, or treatment with therapeutic oral or IV antibiotics within 14 days prior to Day 1 of Cycle 1
* Prior treatment with any KRAS G12C inhibitor or pan-KRAS/RAS inhibitor
* More than 30 Gy of radiotherapy to the lung within 6 months of randomization
* Uncontrolled tumor-related pain
* Unresolved toxicities from prior anticancer therapy
* History of malignancy within 5 years prior to screening, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, nonmelanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 4 years
  PFS is defined as the time from randomization to the first occurrence of disease progression, as determined by blinded independent central review (BICR) according to RECIST v1.1, or death from any cause (whichever occurs first)

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 4 years
  OS is defined as the time from randomization to death from any cause
Confirmed Objective Response | Up to approximately 4 years
  Confirmed objective response is defined as complete response (CR) or partial response (PR) on two occasions ≥ 4 weeks apart, as determined by BICR according to RECIST v1.1
Time to Confirmed Deterioration (TTCD) on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Dyspnea Item and Physical Functioning Scale | Baseline up to approximately 4 years
TTCD on the EORTC Quality-of-Life Questionnaire-Supplemental Lung Cancer Module (QLQ-LC13) Cough Scale | Baseline up to approximately 4 years
Duration of Response (DOR) | Up to approximately 4 years
  DOR is defined as the time from the first occurrence of a documented confirmed objective response to disease progression, as determined by BICR according to RECIST v1.1, or death from any cause (whichever occurs first)
Percentage of Participants with Adverse Events (AEs) | Up to approximately 4 years
Number of Participants Reporting Presence, Frequency, Severity, and/or Degree of Interference with Daily Function of Symptomatic Treatment Toxicities Assessed by NCI Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to approximately 4 years
Change from Baseline in Diarrhea, Nausea, Vomiting, Anorexia, Alopecia, Dyspnea, Cough, Constipation, Myalgia, Headache, and Rash/Acne as Assessed Through use of the NCI PRO-CTCAE | Baseline up to approximately 4 years
Frequency of Participants' Response of the Degree they are Troubled with Treatment Symptoms, as Assessed Through use of the single-item EORTC Item List (IL46) | Up to approximately 4 years
Change from Baseline in Cough, Chest Pain, Dyspnea, Physical and Role Functioning, and Global Health Status score/Quality of Life Score (GHS/QoL) at Each Timepoint as Assessed Through use of the EORTC QLQ-LC13 and QLQ-C30 | Baseline up to approximately 4 years
TTCD on the EORTC QLQ-C30 Role Functioning and GHS/QoL scales | Up to approximately 4 years
TTCD on the Chest Pain Scale of the QLQ-LC13 Scales | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (151):
- United States (25):
  - Banner Health MD Anderson AZ, Gilbert, Arizona
  - Los Angeles Cancer Network, Los Angeles, California
  - UCLA Hematology / Oncology Clinic, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Florida Cancer Specialists - North;725 6th Ave South (St. Petersburg), St. Petersburg, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - New England Cancer Specialists, Westbrook, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Minnesota Oncology Edina, Edina, Minnesota
  - Columbia University Medical Center, New York, New York
  - Taylor Cancer Research Center, Maumee, Ohio
  - Oncology Associates of Oregon, P.C, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC - Chattanooga, Chattanooga, Tennessee
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - JPS Health Network, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Northeast Texas, Longview, Texas
- Argentina (2):
  - Hospital Britanico, Buenos Aires
  - Centro Oncologico Korben, Ciudad Autonoma Buenos Aires
- Australia (5):
  - Liverpool Hospital, Liverpool, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- Krankenhaus Nord - Klinik Floridsdorf, Vienna, Austria
- Belgium (10):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - CHU de Liège (Sart Tilman), Liège
  - CHU UCL Mont-Godinne, Mont-godinne
  - AZ Delta (Campus Rumbeke), Roeselare
  - Vitaz, Sint-Niklaas
  - ZAS Sint Augustinus Wilrijk, Wilrijk
- Brazil (5):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
- Canada (2):
  - William Osler Health Centre - Brampton Civic Hospital, Brampton, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus N
  - Herlev Hospital, Herlev
  - Regionshospitalet Gødstrup, Herning
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio Uni Hospital, Kuopio
- France (12):
  - CHRU Brest, Brest
  - Chu Toulouse, Bron
  - Hopital Louis Pradel, Bron
  - CHRU Lille, Lille
  - Centre Leon Berard, Lyon
  - CHU Montpellier, Montpellier
  - Centre Antoine Lacassagne Centre Régional de Lutte Contre Le Cancer, Nice
  - Hopital Tenon, Paris
  - CHU Bordeaux, Pessac
  - CH de Saint Quentin, Saint-Quentin
  - Chru de Strasbourg, Strasbourg
  - Hia Sainte Anne, Toulon
- Germany (17):
  - Evangelische Lungenklinik Berlin, Berlin
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - Klinikum Koeln-Merheim, Cologne
  - KEM/Evang. Kliniken Essen Mitte gGmbH, Essen
  - Universitätsklinikum Essen, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Asklepios Fachkliniken GmbH, Gauting
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Universität Des Saarlandes, Homburg
  - SLK Kliniken Heilbronn GmbH, Standort Fachklinik Löwenstein, Löwenstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum Bogenhausen, München
  - Universitätsklinikum Münster, Medizinische Klinik A, Translationale Onkologie, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Klinikum Würzburg Mitte gGmbH, Würzburg
- Greece (5):
  - Uoa Sotiria Hospital, Athens
  - Errikos Dynan Hospital, Athens
  - University Hospital of Larissa, Larissa
  - Theageneio Hospital, Thessaloniki
  - Ag. Loukas Hospital, Thessaloniki
- Hong Kong (2):
  - Tuen Mun Hospital, Hong Kong
  - Prince of Wales Hosp, Shatin
- Italy (8):
  - Irccs Ist. Tumori Giovanni Paolo Ii, Bari, Apulia
  - A.O. Universitaria Di Parma, Parma, Emilia-Romagna
  - IRCCS Istituto Regina Elena (IFO), Rome, Lazio
  - Ospedale Policlinico San Martino, Genoa, Liguria
  - Ospedale Civile SS Annunziata, Sassari, Sardinia
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV), Padua, Veneto
- Japan (6):
  - Kyushu University Hospital, Fukuoka
  - Sendai Kousei Hospital, Miyagi
  - Kindai University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- ARKE Estudios Clínicos S.A. de C.V., Mexico City, Mexico
- Netherlands (6):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Ziekenhuis Rijnstate, Arnhem
  - Amphia Ziekenhuis, Breda
  - Ziekenhuis St. Jansdal, Harderwijk
  - Medisch Centrum Haaglanden, locatie Antoniushove, Leidschendam
  - Isala, Zwolle
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Instytut Gruzlicy I Chorob Pluc, Warsaw
  - Dolno?L?Skie Centrum Onkologii, Pulmonologii I Hematologii, Wroc?aw
- Portugal (5):
  - Hospital de Braga, Braga
  - CHUC - Unidade de Pneumologia Oncológica, Coimbra
  - Centro Clinico Champalimaud, Lisbon
  - Centro Hospitalar do Porto ? Hospital de Santo António, Porto
  - IPO do Porto, Porto
- National Cancer Centre, Singapore, Singapore
- South Korea (6):
  - St. Vincent's Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Institut Catala d Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Nuestra Senora de Valme, Seville, Sevilla
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario la Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Gävle Sjukhus, Gävle, Sweden
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Thailand (3):
  - Vajira Hospital, Bangkok
  - Siriraj Hospital - Chulabhorn Bone Marrow Transplant Centre, Bangkok
  - Songklanagarind Hospital, Songkhla
- United Kingdom (9):
  - Addenbrooke's Hospital, Cambridge
  - Castle Hill Hospital, Cottingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James University Hospital, Leeds
  - Guy's Hospital - Cancer Centre, London
  - Royal Marsden Hospital - London, London
  - Nottingham City Hospital, Nottingham
  - Royal Marsden Hospital (Sutton), Sutton
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing